CLINICAL TRIAL: NCT07296133
Title: Evaluating Online Gameplay Intervention to Support Social Engagement in Older Adults With and Without Mild Cognitive Impairment (MCI)
Brief Title: GAMES Intervention in MCI (Mild Cognitive Impairment)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Kayci Vickers, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025P011653; 1R44AG078009-01 (NIH)
Record Dates: First submitted 2025-12-18; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online Gameplay Intervention Group (Experimental): Participants will receive:
  * brief (< 10 minutes) psychoeducation about the importance of engaging in social activities to support cognitive stimulation and brain health
  * technology session to show them how to access games via OneClick
  * participants will receive weekly calls from study staff to provide support and briefly query about social activities that week.
  * A subset of questionnaires will be re-administered after 6 weeks of the intervention to capture any change occurring at intervention mid-point.
  * Following completion of the 12-week intervention, participants will repeat a subset of baseline questionnaires to evaluate for change over time.
  Interventions: Behavioral: Online Gameplay Intervention
- Wait-list control Group (Other): Participants will receive:
  * brief (< 10 minutes) psychoeducation about the importance of engaging in social activities to support cognitive stimulation and brain health
  * Participants will be notified that study team will receive weekly phone calls to ask about social activities they completed in the week prior.
  * Following completion of the 12-week waitlist period, participants will repeat the baseline questionnaires to evaluate for change over time.
  * After completing the waitlist condition, they will be offered the opportunity to complete the gameplay intervention.
  Interventions: Behavioral: Waitlist control

INTERVENTIONS:
Behavioral: Online Gameplay Intervention — -The online gameplay intervention includes playing online versions of common games (such as Connect 4 and Uno) with a partner, 3 times per week for at least 15 minutes, for 12 weeks.
  All games will be delivered via a novel online platform (OneClick; developed by PotLuck, LLC) created specifically to support and enhance social engagement with family members and close friends.
  * Participants will receive weekly calls from study staff to provide support and briefly query about social activities that week.
  * They will not receive reminders or be contacted by the study outside of the weekly phone calls, apart from mid intervention questionnaires.
  Arms: Online Gameplay Intervention Group
Behavioral: Waitlist control — - Participants will be informed that study team will contact them once per week by telephone for 12 weeks, to ask about social activities they completed in the week prior.
  Arms: Wait-list control Group

SUMMARY:
The objective of the present study is to evaluate whether online, remote gameplay can facilitate social engagement and reduce feelings of loneliness and isolation in adults with and without mild cognitive impairment (MCI).

DETAILED DESCRIPTION:
In this study, the investigators will complete a low burden gameplay intervention wherein individuals with and without MCI will be asked to play specially created online versions of common games (such as Connect 4 and Uno) 3 times per week for 12 weeks. Each gameplay session will last at least 15 minutes. Individuals in the intervention condition will begin gameplay immediately, those in the waitlist control condition will complete a 12-week waiting period before beginning gameplay. All games will be delivered via a novel online platform (OneClick; developed by PotLuck, LLC) created specifically to support and enhance social engagement with family members and close friends. In addition to weekly gameplay, participants will receive weekly calls from study staff, both during the waitlist and intervention conditions, to provide support and briefly query about social activities that week. They will also complete a series of questionnaires at 0-, 6-, and 12-weeks of the intervention to evaluate outcomes. The long-term goal of this research is to benefit health and quality-of-life outcomes by delivering remote socialization options to older adults with MCI. OneClick is an easy-to-use platform that has been designed with and for older adults, including those with MCI, to accommodate their unique socialization needs and technology design requirements. The OneClick platform and games used in this study are owned by PotLuck, LLC and therefore stand to be commercialized by their team. Data will not be submitted to the FDA and procedures will not be tested clinically as part of this protocol. In this phase of the study, we will test whether online games delivered via the OneClick platform improve research participants' report of social engagement, isolation, and loneliness alongside other aspects of wellbeing.

ELIGIBILITY:
Inclusion Criteria:

* 50 to 85 years old
* Living independently (note: can live in assisted living, but must have independently complete daily activities)
* Fluent in English
* Adequate visual and auditory acuity to see/hear computer screen
* MoCA-Blind (converted to MoCA score) > 17

Additional Criteria for MCI Group:

* Existing diagnosis by HC professional
* MoCA-Blind (converted to MoCA score) of 18-25
* FAQ < 9

Exclusion Criteria:

* Cognitive impairment secondary to stroke, TBI or other neurological cause without concern for neurodegenerative condition (e.g., Alzheimer's disease, vascular dementia, etc.)
* Medical illnesses that would prevent participation
* Major psychiatric disturbance meeting DSM V criteria in last year
* Hx of substance abuse within last two years
* Current psychoactive med use

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2025-12-08 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Change in friendship Scale score | Pre-intervention (Baseline), week 6 and post-intervention (week 12)
  The scale consists of 5 core items, each with a 5-point frequency response (Almost always to Not at all).
  Total possible score range is 5-25. Higher scores indicate greater feelings of social isolation (worse study outcome).
Change in UCLA Loneliness Scale score | Pre-intervention (Baseline), week 6 and post-intervention (week 12)
  This is a self -report scale with 20 items. Participants rate each item on a 4-point Likert scale:
  (1 = Never, 2 = Rarely, 3 = Sometimes, 4 = Often). Total possible score ranges from 20 to 80, with higher scores indicating greater perceived loneliness (worse study outcome).
Change in Neuro-QOL score | Pre-intervention (Baseline), week 6 and post-intervention (week 12)
  Neuro-QOL ("Quality of Life in Neurological Disorders") consists of a scale designed to measure health-related quality of life across a variety of neurological conditions. The abbreviated form comprises short forms (8-10 items each) covering 13 key domains: physical, mental, and social health. Response format for each item ranges from "Never" to "Always" or severity levels like "None" to "Cannot do". Scores are summarized and represented with T-scores (mean = 50, SD = 10), derived from their respective calibrated item questionnaire. Higher scores correlate with worse outcome.
Change in meaning and purpose score | Pre-intervention (Baseline), week 6 and post-intervention (week 12)
  This scale measures an individual's sense of meaning, purpose, and life satisfaction. Includes 8-9 items in the short form, with statements like "My life has meaning" or "I have a sense of purpose," rated on a 5-point (from 1=never to 5=always). Scores are expressed as T-scores (mean = 50, SD = 10). Higher scores represent better outcome (more positive well-being).

SECONDARY OUTCOMES:
Change in Tech Experience and Comfort scale score | Pre-intervention (Baseline), week 6 and post-intervention (week 12)
  Measures confidence in using new or everyday technologies, reflecting both comfort and perceived ability. Includes 10 items, each beginning with the stem "I could use the new technology…".
  Participant will rate confidence on a 10-point scale (e.g., from "Not at all confident" to "Completely confident"). Total possible score range is 10-100, with better score correlating with greater confidence/comfort in using technology.
Change in Perceived Stress score | Pre-intervention (Baseline), week 6 and post-intervention (week 12)
  Measures the degree to which situations in one's life are appraised as stressful.
  This is a 10-item scale that focuses on feelings of unpredictability, lack of control, and overload during the past month. Response format is with a 5-point Likert scale (0 = Never, 1 = Almost never, 2 = Sometimes, 3 = Fairly often, 4 = Very often). Total score range is 0-40. Higher scores correlate with greater perceived stress (worse outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Kayci Vickers, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlies results reported in as outcomes in publication of RCT results, after being de-identified (includes tables, graphs, appendices, etc.)
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available within 3 months of acceptance for publication and will end 5 years after initial publication.
Access Criteria: Data will be shared with researchers who provide a methodologically sound proposal, to achieve aims in approved proposal.
  Proposals should be directed to kvicker@emory.edu. To gain access, data requestors will need to sign a data access agreement. Data will be made available for 5 years.